CLINICAL TRIAL: NCT06474897
Title: Comparison of the Efficacy of Mulligan Mobilization and Ozone Therapy in Patients With Subacromial Impingement Syndrome
Brief Title: Comparison of Mobilization and Ozone Therapy in Impingement Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Firat University (Other)
Responsible Party: Principal Investigator, Songül Bağlan Yentür, Head of Physiotherapy and Rehabilitation Department, Firat University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024/06-38
Record Dates: First submitted 2024-06-20; First posted 2024-06-26 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Impingement Syndrome
Keywords: Impingement Syndrome; Ozone therapy; Mulligan mobilization

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ozone therapy group (Experimental): Ozone therapy will be practiced to study group. Inject 10 ml of ozone gas (O2-O3) at a concentration of 10 µg/ml 3 times at one week intervals. All injections will be performed by the same experienced specialist doctor.
  Interventions: Other: Ozone therapy
- Mobilization group (Experimental): Mulligan mobilization will be practiced to control group. Mobilizations will be performed once a week for 3 consecutive weeks. The first one is a seated position with the patient's arm in approximately 90° abduction. The patient will be asked to abduct the arm and at the same time the physiotherapist will perform posterio/lateral gliding of the shoulder head with the left hand.
  Interventions: Other: Mulligan Mobilization

INTERVENTIONS:
Other: Ozone therapy — Ozone therapy will be practiced to study group. Inject 10 ml of ozone gas (O2-O3) at a concentration of 10 µg/ml 3 times at one week intervals. All injections will be performed by the same experienced specialist doctor.
  Arms: Ozone therapy group
Other: Mulligan Mobilization — Mulligan mobilization will be practiced to control group. Mobilizations will be performed once a week for 3 consecutive weeks. The first one is a seated position with the patient's arm in approximately 90° abduction. The patient will be asked to abduct the arm and at the same time the physiotherapist will perform posterio/lateral gliding of the shoulder head with the left hand.
  Arms: Mobilization group

SUMMARY:
Studies investigating the efficacy of the Mulligan technique and ozone therapy in patients with shoulder impingement syndrome are limited in the literature. The aim of this study was to compare the effectiveness of Mulligan mobilization method and ozone therapy in patients with shoulder impingement syndrome. Ozone therapy will be practiced to study group. Mulligan mobilization will be practiced to control group. Pain, range of motion and function will be assessed before and after treatment.

DETAILED DESCRIPTION:
The subacromial bursa and rotator cuff muscles are compressed between the acromion and the proximal humerus. If the subacromial surface volume decreases, degeneration and tears of the soft structures may occur during forward extension and rotation. Studies investigating the efficacy of the Mulligan technique and ozone therapy in patients with shoulder impingement syndrome are limited in the literature. The aim of this study was to compare the effectiveness of Mulligan mobilization method and ozone therapy in patients with shoulder impingement syndrome. Ozone therapy will be practiced to study group. Inject 10 ml of ozone gas (O2-O3) at a concentration of 10 µg/ml 3 times at one week intervals. All injections will be performed by the same experienced specialist doctor. Mulligan mobilization will be practiced to control group. Mobilizations will be performed once a week for 3 consecutive weeks. The first one is a seated position with the patient's arm in approximately 90° abduction. The patient will be asked to abduct the arm and at the same time the physiotherapist will perform posterio/lateral gliding of the shoulder head with the left hand. Pain, range of motion and function will be assessed before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 8-65 years
* Patients with shoulder impingement syndrome

Exclusion Criteria:

* Shoulder surgery
* History of scoliosis
* Infection
* Cardiac pacemaker
* Recent myocardial infarction
* Malignancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-06-21 (Estimated); Primary Completion 2024-08-20 (Estimated); Study Completion 2024-09-20 (Estimated)

PRIMARY OUTCOMES:
Pain assessment | 1 minute
  The Visual Analog Scale (VAS), which quantifies parameter values that cannot be measured numerically, will be used to assess the pain intensity of the participants. VAS is a simple and commonly used scale that numerically indicates the severity of pain. A 10 cm line is divided into 10 equal parts and numbered from 0 to 10. The two extremes are defined as the minimum and maximum pain intensity.

SECONDARY OUTCOMES:
Range of motion assessment | 1 minute
  n order to evaluate the active and passive range of motion of the participants, measurements will be made with a goniometer, which gives an objective and numerical value.
Function assessment | 2 minutes
  The Shoulder Arm and Hand Problems Questionnaire (DASH) will be used to assess shoulder function. It is one of the most validated questionnaires used to assess functionality after upper extremity injuries.

CONTACTS AND LOCATIONS:
Locations (1):
- Songul Baglan Yentur, Elâzığ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No